CLINICAL TRIAL: NCT05643547
Title: Immunophenotypic Evaluation of IL-7R α in Acute Leukaemia
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Rania Abdeltwab Abdelazeim (Other)
Responsible Party: Sponsor-Investigator, Rania Abdeltwab Abdelazeim, Immunophenotypic evaluation of IL-7R α in Acute leukaemia, Assiut University
Organization: Assiut University (Other)
Other Study IDs: 159159
Record Dates: First submitted 2022-11-30; First posted 2022-12-08 (Actual); Last update posted 2022-12-08 (Actual); Status verified 2022-11

CONDITIONS: Benefit: To Patient Have Investigation for Diagnosis and Follow up for His Disease and Reach to New Method Help in Early Diagnosis of Lymphoid Disorder

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional

SUMMARY:
Acute leukemia is generally understood to be a neoplastic process that exerts a maturational block at a hematopoietic precursor cell level, accompanied by a proliferative drive of varying degree. The resulting accumulation of cells, most frequently in the marrow, causes the typical clinical picture, which includes marrow failure, tissue infiltration, organomegaly and on occasion, tumor masses. AL is broadly classified as acute myeloid leukemia (AML) and acute lymphoid leukemia (ALL) (1).

Acute lymphoblastic leukemia is frequently diagnosed in children and young adults, with incidence peaks between 2 and 5 years of age (2), whereas AML is the most common acute type in adults (3).

In addition to leukemia cells themselves, cells of the immune system are a fundamental component of the tumor microenvironment (TME), which often modify the TME to be more favorable to tumor development and progression through producing cytokines and mediators (4,5) . Interleukins / interleukin receptors interaction plays important roles in the antitumor immune response through mediating cell-cell communication in TME and is reported to be relevant to patient prognosis (6,7). As a member of the Interleukin family, Interleukin 7 (IL7) play vital roles in hematopoiesis and the development of T lymphocytes, as well as the inflammation, autoimmune diseases and hematological cancers. Its function is mediated by the IL7 R, which is a membrane receptor consisted of the specific IL7Ra chain (CD127) and IL-7Rγ chain (common gamma chain shared by the receptors for IL-2,-4,-9,-15, and-21) (8). It is thus not surprising that activation of IL-7 signalling is seen in the majority of T-ALLs and in some of the B cell precursor ALL (9,10).

Consistent with the absolute requirement of IL-7 to human T cell development, most T-ALLs have been shown to respond to IL-7. Thus targeting IL-7 signaling might be a reasonable general approach for treatment of T-ALL, regardless the presence of activating mutations. (10)

DETAILED DESCRIPTION:
Acute leukemia is generally understood to be a neoplastic process that exerts a maturational block at a hematopoietic precursor cell level, accompanied by a proliferative drive of varying degree. The resulting accumulation of cells, most frequently in the marrow, causes the typical clinical picture, which includes marrow failure, tissue infiltration, organomegaly and on occasion, tumor masses. AL is broadly classified as acute myeloid leukemia (AML) and acute lymphoid leukemia (ALL) (1).

Acute lymphoblastic leukemia is frequently diagnosed in children and young adults, with incidence peaks between 2 and 5 years of age (2), whereas AML is the most common acute type in adults (3).

In addition to leukemia cells themselves, cells of the immune system are a fundamental component of the tumor microenvironment (TME), which often modify the TME to be more favorable to tumor development and progression through producing cytokines and mediators (4,5) . Interleukins / interleukin receptors interaction plays important roles in the antitumor immune response through mediating cell-cell communication in TME and is reported to be relevant to patient prognosis (6,7). As a member of the Interleukin family, Interleukin 7 (IL7) play vital roles in hematopoiesis and the development of T lymphocytes, as well as the inflammation, autoimmune diseases and hematological cancers. Its function is mediated by the IL7 R, which is a membrane receptor consisted of the specific IL7Ra chain (CD127) and IL-7Rγ chain (common gamma chain shared by the receptors for IL-2,-4,-9,-15, and-21) (8). It is thus not surprising that activation of IL-7 signalling is seen in the majority of T-ALLs and in some of the B cell precursor ALL (9,10).

Consistent with the absolute requirement of IL-7 to human T cell development, most T-ALLs have been shown to respond to IL-7. Thus targeting IL-7 signaling might be a reasonable general approach for treatment of T-ALL, regardless the presence of activating mutations. (10).

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed patients with Acute leukemia (ALL, AML), male or female at any age.

Exclusion Criteria:

* Patients diagnosed with hematological malignancy other than acute leukemias
* Patients receiving chemo and/or radiotherapy
* Patients on steroid therapy for any other reason
* Patients receiving any immunosuppressive drug

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: - Newly diagnosed patients with Acute leukemia (ALL, AML), male or female at any age will be investigated for Immunophenotypic expression of IL7R α and its diagnostic value.
Sampling Method: Probability Sample
Enrollment: 83 (Estimated)
Dates: Start 2023-03-01 (Estimated); Primary Completion 2023-12-30 (Estimated); Study Completion 2024-10-30 (Estimated)

PRIMARY OUTCOMES:
Immunophenotypic expression of IL7R α in acute leukemia cases. | 2022-2024
  Immunophenotypic expression of IL7R α in acute leukemia cases.